CLINICAL TRIAL: NCT02520856
Title: New Diagnostic Strategy in Hypertrophic Cardiomyopathy Including a New Genetic Approach: A Multicentric Prospective Study
Brief Title: New Diagnostic Strategy in Hypertrophic Cardiomyopathy
Acronym: HYPERGEN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-29; RCAPHM14_0358 (Registry Identifier: Assistance Publique Hôpitaux de Marseille)
Record Dates: First submitted 2015-08-05; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypertrophic cardiomyopathy: All patients with newly diagnosed unexplained HCM will be prospectively included.
  All patients will undergo both classical genetic analysis and WES technology.
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample

SUMMARY:
Hypertrophic cardiomyopathy (HCM) is an autosomal dominant disease characterized by unexplained hypertrophy of the left ventricle, often with predominant involvement of the interventricular septum, and characterized by myocyte disarray and fibrosis.

HCM is the most common familial heart disease with strong genetic heterogeneity, demonstrated over the past 20 years. Mutations in 11 or more genes encoding proteins of the cardiac sarcomere are responsible for (or associated with) HCM.

However, 30-40% of sporadic and familial cases of HCM are still genetically unlabelled. In addition, secondary HCM caused by Fabry's disease or amyloidosis, may mimic primary HCM and may be under diagnosed. This may result in a delay in accurate diagnosis and instauration of specific treatment, with possible clinical consequences for the patients.

For these reasons, we decided to apply a new diagnostic strategy for patients with newly diagnosed HCM, including the whole exome sequencing (WES) technology.

If correctly applied, this new technology has the potential to strongly reduce the diagnostic wavering leading to earlier diagnosis and genetic counseling in sarcomeric HCM and rarer forms of secondary HCM including Fabry's disease and amyloidosis, and also specific therapy set-up in secondary forms of HCM. It should also allow identifying new genes responsible for HCM.

DETAILED DESCRIPTION:
Background : Hypertrophic cardiomyopathy (HCM) is an autosomal dominant disease characterized by unexplained hypertrophy of the left ventricle, often with predominant involvement of the interventricular septum, and characterized by myocyte disarray and fibrosis.

HCM is the most common familial heart disease with strong genetic heterogeneity, demonstrated over the past 20 years. Mutations in 11 or more genes encoding proteins of the cardiac sarcomere are responsible for (or associated with) HCM.

However, 30-40% of sporadic and familial cases of HCM are still genetically unlabelled. In addition, secondary HCM caused by Fabry's disease or amyloidosis, may mimic primary HCM and may be under diagnosed. This may result in a delay in accurate diagnosis and instauration of specific treatment, with possible clinical consequences for the patients.

Objectives : For these reasons, we decided to apply a new diagnostic strategy for patients with newly diagnosed HCM, including the whole exome sequencing (WES) technology.

1. Main objective: to evaluate the additional diagnostic value of the new proposed strategy for the identification of a specific cause of HCM as compared with conventional diagnostic strategy
2. Secondary objectives:

To evaluate the frequency of secondary HCM (Fabry's disease, amyloidosis, mitochondrial cardiomyopathies, and others) observed by this systematic screening in a population of newly diagnosed HCM

Perspectives: If correctly applied, this new technology has the potential to strongly reduce the diagnostic wavering leading to earlier diagnosis and genetic counseling in sarcomeric HCM and rarer forms of secondary HCM including Fabry's disease and amyloidosis, and also specific therapy set-up in secondary forms of HCM. It should also allow identifying new genes responsible for HCM.

ELIGIBILITY:
Inclusion Criteria:

* patient with newly diagnosed hypertrophic cardiomyopathy (HCM), based on conventional echocardiographic criteria.The diagnosis of HCM will be considered definite in the presence of left ventricle hypertrophy without cavity dilatation and without other cardiac or systemic disease able to produce the magnitude of hypertrophy.

Exclusion Criteria:

* Associated cardiac or non cardiac disease known to cause left ventricle hypertrophy (uncontrolled systemic Hypertension, severe aortic stenosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with unexplained Hypertrophic cardiomyopathy will be prospectively included.
  HCM diagnosis will be based on conventional echocardiographic criteria and will be considered definite in the presence of LV hypertrophy without cavity dilatation and without other cardiac or systemic disease able to produce the magnitude of hypertrophy.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
whole exome sequencing | 12 months
Classic genetic analysis | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France